CLINICAL TRIAL: NCT02075216
Title: Transurethral Autologous Myoblast Injection for Treatment of Urinary Incontinence in Children With Bladder Exstrophy
Brief Title: Transurethral Myoblast Injection for Urinary Incontinence in Children With Bladder Exstrophy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Collaborators: Cairo University (Other); Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Sayed Bakry, Associate Professor , Consultant of Isolation and Culturing of Stem Cells, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT1502231; Azhar2013298 (Other: Al Azhar University)
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Children; Bladder Exstrophy; Extrophy -Epispadias complex,; Modern staged repair,; Bladder neck reconstruction
MeSH Terms: conditions — Urinary Incontinence; Bladder Exstrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myoblasts Preparation (Experimental): Myoblast Preparation, Myoblast Transplantation & Neonatal Cystourethroscope Injection
  Approximately 8 to 10 gm muscle will be obtained from the rectus abdominis. Patient muscle fibers will be isolated using the fiber explant technique described by Rosenblatt et al, with some modifications. Culture conditions will be mainly adapted from Rando and Blau.
  After 22 days of culture myoblasts will be harvested by trypsinization and incubated in serum-free medium during the last 2 hours before injection. Immediately before injection the cell pellet will be resuspended in autologous serum and/ or platelet rich plasma (PRP).
  Interventions: Procedure: Myoblast Transplantation; Biological: Neonatal Cystourethroscope Injection

INTERVENTIONS:
Procedure: Myoblast Transplantation — For each patient 4-7 Million cells per ml will be injected into 8 to 10 sites through a cystoscopic injection needle with a 10 mm long, 21 gauge needle connected to a 30 cm long plastic tube, using a 6.75Fr neonatal cystourethroscope. The suspension will be injected in the area of the external sphincter and along the posterior urethra proximal to the verumontanum, aiming to attain visual occlusion of the urethral lumen.
Biological: Neonatal Cystourethroscope Injection — 4-7 Million cells per ml will be injected into 8 to 10 sites through a cystoscopic injection needle with a 10 mm long, 21 gauge needle connected to a 30 cm long plastic tube, using a 6.75Fr neonatal cystourethroscope.

SUMMARY:
Muscle precursor cells constantly regenerate striated muscles, and include the quiescent satellite cells located beneath the basal lamina of skeletal myofibers, which are responsible for repair of the terminally differentiated striated muscle tissue. Transurethral implantation of autologous myoblasts may represent an improved alternative to synthetic bulking agents, with the unique ability to compensate for the deficient muscle fibers in the urethral sphincter. Clinical studies of cell therapy based treatment of sphincter insufficiency, using muscle derived stem cell transplantation was carried out in patients with stress incontinence revealed and confirmed the ability of cell therapy to improve the structure and contractile function of the sphincter. In this study autologous heterotopic myoblasts will be transurethrally injected in patients with bladder extrophy epispadias complex who remained incontinent after staged bladder reconstruction and bladder neck reconstruction.

The aim of this study is to investigate the potential therapeutic effects of autologous myoblast injection for the treatment of children presenting with urinary incontinence after modern staged repair and bladder neck reconstruction of extrophy-epispadias complex as well as studying the safety, efficacy and durability of the procedure, and health related quality of life.

DETAILED DESCRIPTION:
Achieving urinary continence in patients with bladder extrophy epispadias complex remains a challenging urological goal. Children with bladder extrophy epispadias complex generally undergo many surgical procedures for the treatment of sphincteric incompetence, including bladder neck reconstruction, slings and bulking agent injection. The key point in most of these procedures is to enhance urethral resistance, leading to some degree of bladder outlet obstruction. However, the reported 7% to 85% continence rates in these patients may not exactly represent those children who achieve volitional voiding through the urethra, but may also include the ones with bladder augmentation and urinary diversion. Endoscopic injection of bulking agent has emerged as a therapeutic approach in the treatment of urinary incontinence (UI). this procedure seems to be economical, with shorter hospitalization and fewer major complications. On the other hand, degradation, migration, reabsorption, overbulking, bladder outlet obstruction and hypersensitivity are frequently reported complications of bulking agents.

The ideal substance for periurethral injection should be durable, non immunogenic, nonmigratory and efficacious. So, transurethral implantation of autologous myoblasts may represent an improved alternative to synthetic bulking agents, with the unique ability to compensate for the deficient muscle fibers in the urethral sphincter. Patients with incontinence usually have decreased resting tone and contractility of the rhabdosphincter. In patients with bladder extrophy epispadias complex the perineal structures are dislocated laterally, and the internal and external urethral sphincters are deficient. Muscle precursor cells constantly regenerate striated muscles, and include the quiescent satellite cells located beneath the basal lamina of skeletal myofibers, which are responsible for repair of the terminally differentiated striated muscle tissue. After injury or in response to intensive physical exercise satellite cells proliferate and differentiate into myoblasts, which ultimately fuse to form new myofibers capable of muscle contraction. Considering the limited capacity of the rhabdosphincter for regeneration, the idea of urethral sphincter repair in patients with bladder extrophy epispadias COMPLEX via transurethral injection of autologous myoblasts has been suggested. The technical availability of these cells, as well as immunological acceptance and survival, makes them appropriate for this purpose. Satellite cells are committed cell lineage with restricted plasticity and do not multiply beyond the required repair needs. This property confers an acceptable measure of safety for clinical applications. The first clinical study of cell therapy based treatment of sphincter insufficiency, using muscle derived stem cell transplantation was carried out in patients with stress incontinence revealed and confirmed the ability of cell therapy to improve the structure and contractile function of the sphincter.

ELIGIBILITY:
Inclusion Criteria:

Gender: male.

Ages: above 2 Years old.

Patient with Urinary incontinence after successful staged repair and bladder neck reconstruction of extrophy -epispadias complex.

Absence of urinary tract infection after urine analysis and urine culture.

Serum creatinine in normal range for age.

Parent or legal guardian agrees to complete and sign the informed consent document.

-

Exclusion Criteria:

Any degree of Spinal cord injury, systemic, neuronal paralysis or sacral agenesis.

Urodynamic study demonstrating severe uninhibited bladder contractions.

Severe urethral or bladder neck stricture demonstrated during screening cystoscopy or cystogram

Cystography at the time of screening demonstrating Grade IV vesicoureteral reflux (high-grade reflux with dilation of the renal pelvis and blunting or the fornices) or Grade V vesicoureteral reflux (Grade IV findings plus loss of the papillary impression and ureteral tortuosity).

Any degree of renal scarring at the time of screening as demonstrated by DMSA or MAG3 renal scintigraphy in the presence of any grade of vesicoureteral reflux (VUR)

Renal ultrasound demonstrating Society of Fetal Urology Grade III hydronephrosis (widely split renal pelvis, renal calices uniformly dilated, no parenchymal thinning) or Grade IV hydronephrosis (Grade III dilation plus parenchymal thinning).

Positive urine culture resistant to preoperative oral antibiotic therapy. Immunocompromise patient.

Previous adverse reaction to anesthesia

-

Ages: 2 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Parameters | 12 Weeks
  Clinical assessment.
  Assessment of Continent Score.
  Maximum dry interval per day.

SECONDARY OUTCOMES:
Clinical Changes In Bladder Behavior | 24 Weeks
  Urodynamic Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Wahab El-Okby, MD, Principal Investigator — Deaprtment of Pediatric Surgery School of Medicine Al Azhar University; Abd-Elmoneim Shawky Shams El-deen, MD, Study Chair — Department of Pediatric Surgery , School of Medicine, Al Azhar University; Hussein Galal, MD, Study Chair — Department of Urology, School of Medicine, Al Azhar University; Sayed Bakry, PhD, Study Director — Laboratory of Molecular Biology , School of Science, Al Azhar University; Hala Gabr, MD, Study Chair — Department of Clinical Pathology , School of Medicine, Al Azhar University; Wael Abu El Khier, MD, Study Chair — Department of Clinical Pathology and Immunology, Military Academy; Ahmed Said Sayed Bayomy, MSc, Study Chair — Department of Pediatric Surgery, School of Medicine, Al Azhar University
Locations (1):
- Pediatric Surgery Outpatients Clinics - Al Hussien Hospital, Madīnat an Naşr, Cairo Governorate, Egypt